CLINICAL TRIAL: NCT06350955
Title: Intravenous Iron-induced Hypophosphatemia in Patients With Roux-en-Y Gastric Bypass: a Single-blind, Randomized Clinical Trial Comparing Iron Isomaltoside (Monofer®) and Ferric Carboxymaltose (Ferinject®)
Brief Title: IV Iron-induced Hypophosphatemia After RYGB
Acronym: IVORY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lucie Favre (Other)
Responsible Party: Sponsor-Investigator, Lucie Favre, Co-director of the Obesity Center, CHUV, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-01389
Record Dates: First submitted 2024-03-28; First posted 2024-04-08 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hypophosphatemia; Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Hypophosphatemia | interventions — iron isomaltoside 1000; ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients with Roux-en-Y gastric bypass and iron deficiency 1 (Experimental)
  Interventions: Drug: Iron isomaltoside
- Patients with Roux-en-Y gastric bypass and iron deficiency 2 (Experimental)
  Interventions: Drug: Iron Carboxymaltose

INTERVENTIONS:
Drug: Iron isomaltoside — single dose of 500 mg iron isomaltoside
  Arms: Patients with Roux-en-Y gastric bypass and iron deficiency 1
Drug: Iron Carboxymaltose — single dose of 500 mg ferric carboxymaltose
  Arms: Patients with Roux-en-Y gastric bypass and iron deficiency 2

SUMMARY:
The primary objective of the study is to compare the incidence of hypophosphatemia in RYGB patients treated with intravenous (IV) single dose of iron isomaltoside (Monofer®) or ferric carboxymaltose (Ferinject®).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Signed informed consent
* Patients with previous RYGB surgery performed > 12 months ago
* Failed response to oral iron supplementation
* Established diagnosis of iron deficiency by ferritin < 50 ug/l or serum ferritin ≤100ug/l and low transferrin saturation (TSAT) ≤ 30%
* Normal phosphate blood level (0.8 - 1.45 mmol/l) before infusion
* Normal magnesium blood level (0.65-1.05 mmol/l)
* Outpatient

Exclusion Criteria:

* - Patients with known hypersensitivity to iron preparation and/or anaphylaxis from any cause
* Patients for whom a treatment with one of the IV iron is contra-indicated (based on product summary of product characteristics)
* Women who are pregnant or breastfeeding
* Intention to become pregnant during the course of the study
* Renal failure, chronic kidney disease stage 3b or worse (eGFR ≤ 45 ml/min/1.73m2)
* Patients who received IV iron infusion during the last 3 months before screening
* Treatment with erythropoietin or erythropoietin-stimulation agents, red blood cell transfusion within the last 3 months prior to screening
* Alcohol or drug abuse within the past 6 months
* Planned surgical procedure within the clinical trial period
* Surgery under general anaesthesia within the last 3 months prior to screening
* Hyperparathyroidism
* Kidney transplantation
* Inability to follow study procedures or give informed consent
* Use and inability to stop from V0 to study end, phosphate supplementation (except daily multivitamin preparation recommended after bariatric surgery; the exact amount of phosphate and iron supplementation in the daily multivitamin will be recorded)
* Osteoporosis drug therapy (bisphosphonates, denosumab or selective oestrogen receptor modulators).
* Patient who refuses to be informed of incidental discoveries that may contribute to the prevention, diagnosis, and treatment of existing or probable future illnesses.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
incidence of hypophosphatemia in RYGB patients treated with intravenous iron | day 14 ± 2, 21 ± 2 and 28 ± 2

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland